CLINICAL TRIAL: NCT04653870
Title: Comparison the Effect of Cyriax Manipulation and Decompression in Patient With Lumber Disc Protrusion
Brief Title: Comparison of Cyriax Manipulation and Decompression in LDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/00681 Salma Bibi
Record Dates: First submitted 2020-11-28; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Lumbar Disc Herniation
Keywords: Herniation; Cyriax manipulation; decompression; bulge; protruded; extruded
MeSH Terms: conditions — Intervertebral Disc Displacement; Hernia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cyriax manipulation (Experimental): cyriax manipulation have three types of classes, rotation, extension and anti-deviation, which is further divided into subclasses. On the inferior level of lumber spine L4-L5 and L5-S1rotation intervention of manipulation are capable of having striking effects of decreasing herniation. First of all we have to perform the simple 'stretch' on lumber spine, which is being the little rotation pressure applied on the body. The patient position of the body is in side lying with the effected side upward so that the outside part of the joint are separated easily on the involved side. After that, whenever it is essential by making use of femur as a rigid bar or support, this maneuver is go along with powerful rotation technique.
  Interventions: Other: cyriax manipulation lumber
- lumber decompresion (Experimental): Spinal decompression therapy has been developed a treatment without surgery for the prolapsed disc and deteriorative spinal disc disease one of the considerable reason for low back pain. This noninvasive interventional treatment for herniated disc and deteriorative disc diseases operated on the principle of remarkably decreasing the pressure on the disc between vertebras.
  Interventions: Other: lumber decompression

INTERVENTIONS:
Other: cyriax manipulation lumber — In group A patients were treated with conservative therapy (hot pack, Kaltenborn soft tissue techniques and home plan) and Cyriax manipulation.
  Exercises (Guided low back exercises, 3-5times/day). Ankle pumping (5-10 repetition with 15-20 second hold), Quads Isometric (5-10 repetition with 15-20 second hold), Hams & Calf stretching (5-10 repetition with 15-20 second hold), Bridging (5-10 repetition with 15-20 second hold), Prone Back extension (10 repetition) Precaution Prevent yourself from sitting low on ground, Sitting with support will be directed and be careful during driving and ascending stairs.
  Cyriax Manipulation: 2-3 repetitions/session, 2 session/week Lumbar spinal manipulation Rotation Techniques Lumbar spinal manipulation Extension Techniques Lumbar spinal manipulation Antideviation Techniques total of 4 session were given. 2 session/week.
  Arms: cyriax manipulation
Other: lumber decompression — Group B: In group B patients were treated with conservative therapy (hot pack, Kaltenborn soft tissue techniques and home plan) and Decompression Session.
  Conservative therapy: Same as Group A
  Lumbar spine decompression:
  30 Minutes Session (generalized time for every one) . On the account of MRI description level is recommended and acknowledged by MRI the level of disc protrusion, decompression is operated. Patient is lying on table facing upward. For locking of the patient's body it was secured by pelvis and thoracic straps. One part of the decompression table is immobile other is movable. Bottom extreme part of the table is mobile.
  Estimation of weight of patient is first thing to do. We calculated it by division of whole weight by 5 and that 5th segment of weight was utilized as an interventional pound for decompression. .
  Arms: lumber decompresion

SUMMARY:
In this study, compare the effects of Cyriax manipulation and Decompression in patient with lumber disc prolapseThis research will provide an important addition to the evidence based treatment intervention in physical therapy in the field of manipulation as there is no such research work have been done on comparative study of cyriax manipulation and decompression in lumber disc protrusion.

DETAILED DESCRIPTION:
According to an estimate, 70 to 80% of the adult population will experience a clinically relevant episode of LBP at some time in their lives. Within the vast differential of LBP, the most common source is intervertebral degeneration leading to degenerative disc disease and LDH. The efficacy of manipulative physical therapy, physical therapy intervention and therapy by general practitioner (GP) for persistent general LBP and neck pain was investigated on 256 patients how didn't received any of the above therapy in last two years were contained in this study. Physical therapy included workout exercises, massage, and physical therapy (related to hot pack, different pain modalities like therapeutic ultrasound, shortwave diathermy, and electrotherapy). Manual therapy includes manual reduction by manipulation and mobilization of the back. Interventions received by GP is medicine related (different types of pain killer and muscles relaxant), guidance about the posture, home plan exercises and different healthy activities and proper rest. Placebo intervention included adjustable shortwave diathermy session for (10 minutes), and adjusted therapeutic ultrasound session for (10 minutes). Recovery rate in the leading complaint was increased with the group receiving manual therapy intervention (4.5) as compare to physical therapy (3.8), after a detailed one year of continuous therapy. There is a great progression seen in physical work by manual therapy. Moreover, manipulation is get going improved gradually, as compare to physiotherapy following in period of 12 months.

The first meta-analysis estimated the efficacy of SMT for LBP due to LDH with other therapies come to the result that SMT was equally effective when compare to other traditional therapies. However a past systematic review was come to the conclusion that SMT was secure and effective in relation to its costs for managing SLDD like LDH, that conclusion was quoted to promote by a very few publications.

One of the present research studies after one year of continuation showed decrease in pain and increase in recreational activities to a long period of time, an additional research work in 2016 described, a remarkable progression in sciatica after 30 days, in patients with lumber discs extrusion and sequestration, as a result of HVLA thrust.

In spite of the factor that there is only average numbers of documentation in the written work which promoted the utilization of SMT to manage LDH, it is extensively applied by therapist.

the comparison of cyriax manipulation and decompresion is an important adding to the researches in evidence based practices. there is no such work done before on comparison of both intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients having Lumber disc prolapse of L1-L5 and S1 (both gender)
* Patients having MRI reports of protruded disc

Exclusion Criteria:

* Inflammatory condition( systemic inflammatory disease of spine)
* Spinal diseases (other than Musculoskeletal)
* Severe radiculopathies (bilateral)
* Operated patients (spine)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-08-25 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Inclinometer | 2nd week
  Inclinometer: Dual inclinometer is used to measure dynamic ROM of lumber spine. For measuring the ROM of flexion, extension and side bending to both sides, place one inclinometer on T12 and the other on S1. Ask the patient to bend forward for flexion, bend backward for extension and sideways for side bending. Note both the readings and subtract the lower one from the above.
goniometer | 2nd week
  Goniometer is used to measure SLR range before and after the treatment For the patients to perform SLR, participants lay supine on a table and are asked to actively raise their leg from the table while keeping their knee straight. Reproduction of the patient's characteristic pain or demonstration of weakness can lead to decreased range of SLR. Symptom production between the ranges of 30 degrees to 60 degrees is an indication of disc pathology.
Numeric pain rating scale | 2nd week
  Numeric pain rating scale: Pain is measured by NPRS before Treatment and after treatment. The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the pain where zero is no pain and 10 is maximum pain (for back and leg)
Oswestry disability index (ODI) | 2nd week
  Oswestry disability index (ODI): Disability is measured by ODI before Treatment and after treatment. It is an extremely important tool that researchers and disability evaluators use to measure a patient's permanent functional disability. The test is considered the 'gold standard' of low back functional outcome tools. it consist of 10, five parts sections. at the end,s core is calculated by dividing the obtained score by total 50, and multiplied by 100. as the sexual section is missing due to ethical reason so total score is 45 instead of 50.

CONTACTS AND LOCATIONS:
Overall Officials: Affan Iqbal, Phd*, Principal Investigator — Riphah International University
Locations (1):
- Max health hospital and rehab center G8 islamabad, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kocak FA, Tunc H, Tomruk Sutbeyaz S, Akkus S, Koseoglu BF, Yilmaz E. Comparison of the short-term effects of the conventional motorized traction with non-surgical spinal decompression performed with a DRX9000 device on pain, functionality, depression, and quality of life in patients with low back pain associated with lumbar disc herniation: A single-blind randomized-controlled trial. Turk J Phys Med Rehabil. 2017 Feb 16;64(1):17-27. doi: 10.5606/tftrd.2017.154. eCollection 2018 Mar. PMID 31453485
- [Background] Koes BW, Bouter LM, van Mameren H, Essers AH, Verstegen GM, Hofhuizen DM, Houben JP, Knipschild PG. Randomised clinical trial of manipulative therapy and physiotherapy for persistent back and neck complaints: results of one year follow up. BMJ. 1992 Mar 7;304(6827):601-5. doi: 10.1136/bmj.304.6827.601. PMID 1532760
- [Background] Leemann S, Peterson CK, Schmid C, Anklin B, Humphreys BK. Outcomes of acute and chronic patients with magnetic resonance imaging-confirmed symptomatic lumbar disc herniations receiving high-velocity, low-amplitude, spinal manipulative therapy: a prospective observational cohort study with one-year follow-up. J Manipulative Physiol Ther. 2014 Mar-Apr;37(3):155-63. doi: 10.1016/j.jmpt.2013.12.011. Epub 2014 Mar 11. PMID 24636109
- [Background] Ehrler M, Peterson C, Leemann S, Schmid C, Anklin B, Humphreys BK. Symptomatic, MRI Confirmed, Lumbar Disc Herniations: A Comparison of Outcomes Depending on the Type and Anatomical Axial Location of the Hernia in Patients Treated With High-Velocity, Low-Amplitude Spinal Manipulation. J Manipulative Physiol Ther. 2016 Mar-Apr;39(3):192-9. doi: 10.1016/j.jmpt.2016.02.013. Epub 2016 Mar 28. PMID 27034106
- [Background] Oh H-J, Jeon C-B, Jeong M-G, Choi S-J. The effects of spinal decompression therapy on pain and disability in patients with chronic low back pain. The Journal of Korean Physical Therapy. 2017;29(6):299-302.